CLINICAL TRIAL: NCT03161418
Title: Study of the Safety of KSP Heptapeptide (KSP-910638G) in Humans for the Early Detection of GI Malignancies
Brief Title: Study of the Safety of KSP Heptapeptide (KSP-910638G)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Danielle Kim Turgeon, Professor of Internal Medicine, Medical School, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00126486
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Healthy Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KSP-910638G 0.4 mg subjects 1-3 (Experimental): The first three subjects will receive lyophilized powder reconstituted with 5 mL of 0.9% NaCl, 0.4 mg of KSP-910638G total. For the first three subjects, 3.34 mL of KSP-910638G will be discarded. The 1.66 mL of KSP-910638G remaining in the syringe will be administered by squirting it into the mouth of the subject.
  Interventions: Drug: KSP-910638G, 0.4 mg
- KSP-910638G 1.2 mg subjects 4-25 (Experimental): Following a safety review of the first three subjects receiving 0.4 mg dose, the remaining 22 subjects will receive the full 1.2 mg dose of KSP-910638G reconstituted in 5 mL 0.9% NaCl. These 22 subjects will receive all 5 mL of the peptide solution in a syringe for administration. The agent will not be reconstituted until the subject is ready to squirt the peptide into his or her mouth via syringe. They will be asked to wait 5 minutes and then drink at least 4-8 oz of tap water.
  Interventions: Drug: KSP-910638G, 1.2 mg

INTERVENTIONS:
Drug: KSP-910638G, 0.4 mg — The investigational agent to be used in this study is KSP heptapeptide, which is a fluorescently-labeled peptide composed of a 7-amino acid sequence attached via a 5 amino acid linker to a near-infrared fluorophore, IRDye800CW. (0.4 mg dose)
  Arms: KSP-910638G 0.4 mg subjects 1-3
Drug: KSP-910638G, 1.2 mg — The investigational agent to be used in this study is KSP heptapeptide, which is a fluorescently-labeled peptide composed of a 7-amino acid sequence attached via a 5 amino acid linker to a near-infrared fluorophore, IRDye800CW. (1.2 mg dose)
  Arms: KSP-910638G 1.2 mg subjects 4-25

SUMMARY:
The purpose of this study is to evaluate the safety of orally administered KSP-910638G, a topically administered li-cor IRDye800CW labeled heptapeptide specific for human epithelial growth factor receptor 2 (HER2).

DETAILED DESCRIPTION:
This is a Phase IA study of the safety of an orally administered KSP-910638G heptapeptide for detection of neoplastic tissues in multiple areas of the gastrointestinal tract in humans. The investigators intend to enroll 25 evaluable subjects. The investigators expect to be able to enroll about 1-2 subjects per week, so the study should take about 4-6 months to complete.

Interested, healthy subjects ages 25-100 who respond to recruitment advertising on UMHealthResearch.org and appear to be eligible based responses to inclusion/exclusion criteria questions will be scheduled for a study visit at MCRU. At the study visit, the subjects will review and sign the informed consent and eligibility will be confirmed. If eligible, subjects will provide a blood sample for clinical labs and a urine sample for urinalysis. A negative urine pregnancy test for women of child-bearing potential is required to be eligible. Eligible subjects will consume the reconstituted KSP-910638G. After 5 minutes, subjects will drink a minimum 4-8 ounces of tap water and vital signs will be taken. Subjects will remain in MCRU for observation for 30 minutes. Vital signs will be recorded after 30 minutes. Subjects are required to return to MCRU to have a repeat blood draw for clinical labs and urinalysis within 24 to 48 hours after KSP-910638G ingestion. The study team will conduct a verbal assessment for toxicity at this visit.

ELIGIBILITY:
Inclusion Criteria:

* Not pregnant (willing to have pregnancy test if applicable)
* No recent illness (infection, URI, virus or flu) within 2 weeks,
* Stable health status (i.e. no medication changes within 2 months, no recent surgery, etc. per PI)
* Willing and able to sign informed consent
* Willing and able to drink the peptide and a tap water chaser
* Willing and able to get baseline and 24-48 hours post ingestion labs

Exclusion Criteria:

* Known allergy to li-cor IRDye800CW, a near infrared fluorosphore or derivatives
* Subjects on active chemotherapy or radiation therapy
* Diabetics on insulin/hypoglycemic (due to fasting requirements)

Ages: 25 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Number of subjects with abnormal lab values | 48 hours
  review of laboratory values for abnormalities after intervention with KSP-910638G

CONTACTS AND LOCATIONS:
Overall Officials: Ashley E Cawthon, Study Chair — Michigan Medicine
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States